CLINICAL TRIAL: NCT02707783
Title: Feasibility and Outcomes of Complete Coronary Revascularization Using Bioresorbable Vascular Scaffold in All-comer Patients With Stable and Unstable Angina: A Multi-centre Registry in Russian Population
Brief Title: Feasibility and Outcomes of Complete Coronary Revascularization Using BVS in All-comer Patients With Angina
Acronym: FEASTRU
Status: Completed | Type: Observational
Sponsor: International Foundation for Development of Medical Science and Education Healthy Heart (Other)
Collaborators: KCRI (Other)
Responsible Party: Sponsor
Other Study IDs: FEAST.RU
Record Dates: First submitted 2016-02-18; First posted 2016-03-14 (Estimated); Last update posted 2018-12-13 (Actual); Status verified 2018-08

CONDITIONS: Angina
Keywords: stable and unstable angina; bioresorbable vascular scaffold; BVS; PCI
MeSH Terms: conditions — Angina Pectoris; Angina, Unstable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Bioresorbable vascular scaffold (BVS) implantation: Patients with un/stable angina that require coronary revascularization undergoing the BVS implantation
  Interventions: Device: Bioresorbable vascular scaffold (BVS) implantation

INTERVENTIONS:
Device: Bioresorbable vascular scaffold (BVS) implantation

SUMMARY:
The aim of the study is feasibility of complete coronary revascularization with bioresorbable vascular scaffold (BVS) implantation and assessment of treatment outcomes in a group of consecutive patients with stable and unstable angina in Russian population.

The hypothesis of this registry study: 1) Complete coronary revascularization with BVS implantation will be feasible to perform in at least 70 percent of patient population with stable and unstable angina qualified for revascularization after coronary angiography, 2) Complete revascularization with BVS is as safe and effective as revascularization with standard BMS (Bare Metal Stent BMS/ Drug Eluting Stent DES stent implantation (published literature comparators in matched populations).

Up to 2500 patients will be enrolled in 13 Russian high volume invasive cardiology centres. 12 month clinical observation and 5-year clinical follow-up is expected.

DETAILED DESCRIPTION:
Study design: Data regarding all consecutive patients qualified for revascularization (PCI Percutaneous Coronary Intervention or CABG Coronary Artery Bypass Grafting) will be collected in this prospective study. Information regarding revascularization strategy will be collected as detailed information concerning PCI procedure. In case of PCI with other than BVS stent implantation (BMS or/and metallic DES) information collected in the study will contain at least:

* Reason why BVS was not implanted
* Final result of baseline treatment
* Acute and long-term outcome of treatment (12 month clinical observation); NB. 5-year clinical follow-up is also expected.

The enrollment phase of the registry is not expected to last longer than 12 months.

ELIGIBILITY:
Inclusion Criteria:

Patient characteristics

* Age > 18 years
* Able and willing to give informed consent
* Willing to comply with specified follow-up evaluations
* Clinical manifestation of coronary artery disease: stable angina or unstable angina
* Indications for coronary revascularization

Exclusion Criteria:

Patient characteristics

* Acute Myocardial infarction
* Cardiogenic shock
* Any reason for patient's inability to comply with 12-month double antiplatelet therapy (DAPT)
* Absolute contraindications to DES or BVS implantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stable and unstable angina qualified for revascularization (PCI or CABG) after coronary angiography.
Sampling Method: Non-Probability Sample
Enrollment: 1602 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Angiographic endpoints: assessment of stent implantation final result:stent delivery, technical success (yes/no) | periprocedural
Angiographic endpoints: assessment of stent implantation final result: percentage of residual stenosis (%) | periprocedural
Angiographic endpoints: assessment of stent implantation final result: dissection (yes/no) | periprocedural
Angiographic endpoints: assessment of stent implantation final result: slow-flow (yes/no) | periprocedural
Angiographic endpoints: assessment of stent implantation final result: no-flow (yes/no) | periprocedural
Angiographic endpoints: assessment of stent implantation final result: distal embolization (yes/no) | periprocedural
Angiographic endpoints: assessment of stent implantation final result: side-branch occlusion (yes/no) | periprocedural
Angiographic endpoints: assessment of stent implantation final result: coronary artery perforation (yes/no) | periprocedural
Acute gain (mm) | periprocedural
Major Adverse Cardiovascular Events | From hospital discharge till 12 months follow up
Major Adverse Cardiovascular Events | in 12 month follow up
TVF (Target Vessel Failure) | in 12 month follow-up
Any revascularization | in 12 month follow-up
  Numbers of any revascularization per patient.
Stent thrombosis (possible and probable) | in 12 month follow-up
Periprocedural MI (Myocardial Infarction) (yes/no) | periprocedural
Angina assessment questionnaire | 12 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Musiałek, MD DPhil, Study Chair — John Paul II Hospital in Krakow, Poland
Locations (14):
- Russia (14):
  - Federal Center for Cardiovascular Surgery, Chelyabinsk, Av. Hero of Russia 2 Rodionov E.N.
  - Federal Cardiovascular Center, Krasnoyarsk, Karaulnaya 45
  - Regional Hospital, Magadan, Nagaevskaya 40
  - Regional Clinical Hospital n.a. S.V., Krasnodar, Ochapovskogo
  - Federal Cardiovascular Center, Kaliningrad
  - Federal State Budgetary Scientific Institution Research Institute for Complex Issues of Cardiovascular Diseases, Kemerovo
  - Regional Clinical Hospital, Krasnoyarsk
  - Clinical Hospital No 1 of Department of Presidents Affairs, Moscow
  - President's Hospital with Policlinic, Moscow
  - Central Railway Hospital 2, Moscow
  - CELT Hospital, Moscow
  - City Clinical Hospital named S.S.Yudina Department of Health of the City of Moscow, Moscow
  - Federal Cardiovascular Center, Perm
  - Tyumen Cardiology Center, Tyumen

IPD SHARING:
Plan to Share IPD: Undecided